CLINICAL TRIAL: NCT06585709
Title: The Development and Validation of Neural Targets in Opioid Use Disorder
Brief Title: OUD (Opioid Use Disorder) Target Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00116151
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Active rTMS (Experimental): A total of 30-sessions of standard iTBS (1800 pulses) will be delivered. rTMS-sessions will be ideally administered over 1-week (10-sessions-per-day, 50-minutes inter-session-interval, 5-days), but there will be flexibility in the delivery paradigm so long as participants complete all sessions of rTMS within 6 weeks and come in at least twice per week.
  Interventions: Device: Active repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham rTMS (Sham Comparator): Double-blind sham-rTMS in an identical fashion to the active-rTMS condition will be delivered.
  Interventions: Device: Sham repetitive Transcranial Magnetic Stimulation (rTMS)
- High Ventral Striatal Reactivity (Other): We will test for ventral striatal reactivity using a Reassessment of Craving MRI task and define high ventral striatal reactivity as having >mean voxels in the ventral striatum activate
  Interventions: Diagnostic Test: High Ventral Striatal Reactivity
- Low Ventral Striatal Reactivity (Other): We will test for ventral striatal reactivity using a Reassessment of Craving MRI task and define low ventral striatal reactivity as having < mean voxels in the ventral striatum activate
  Interventions: Diagnostic Test: Low Ventral Striatal Reactivity

INTERVENTIONS:
Device: Active repetitive Transcranial Magnetic Stimulation (rTMS) — Active rTMS will be delivered with a MagVenture MagPro X100 rTMS device with a Cool-B65-AP coil. rTMS will be applied to a personalized treatment target within the Left-Dorsolateral Prefrontal Cortex using a Localite Neuronavigation device.
  Arms: Active rTMS
Device: Sham repetitive Transcranial Magnetic Stimulation (rTMS) — Sham rTMS in an identical fashion to the active-rTMS condition will be delivered via the built-in e-sham system in the MagVenture device.
  Arms: Sham rTMS
Diagnostic Test: High Ventral Striatal Reactivity — We will test for ventral striatal reactivity using a Reassessment of Craving MRI task and define high ventral striatal reactivity as having >mean voxels in the ventral striatum activate
  Arms: High Ventral Striatal Reactivity
Diagnostic Test: Low Ventral Striatal Reactivity — We will test for ventral striatal reactivity using a Reassessment of Craving MRI task and define low ventral striatal reactivity as having <mean voxels in the ventral striatum activate
  Arms: Low Ventral Striatal Reactivity

SUMMARY:
In this research study the investigators will work with 80-participants with opioid use disorder who are starting treatment with the medication buprenorphine and are trying to quit using opioids.

The investigators are trying to learn two things:

1. Can an MRI brain marker be used to predict which participants will be successful in quitting opioids with buprenorphine?
2. Does adjunctive treatment with repetitive Transcranial Magnetic Stimulation (rTMS) help people quit using opioids more than a sham (placebo) version of rTMS?

In order to complete the study the investigators will ask participants to:

* Complete an MRI within 5-days of starting buprenorphine and again after they are on a full stable dose 1-3 weeks later.
* Undergo study-treatment with 30-sessions of either real or placebo rTMS in as little as 1-week (10-sessions-per-day for five days) or as long as over 6-weeks.
* Meet with the investigators once per week over the following 12-weeks to see if the participants have been able to quit using opioids over that time.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older; all genders included.
2. Intellectual level sufficient to provide informed consent and accurately complete assessment instruments (English speaking/writing).
3. Meet DSM-5 criteria for moderate or severe OUD. Individuals may also meet criteria for another substance use disorder (with the exception of alcohol or sedative/hypnotic); but must identify opioids as their primary substance.
4. Starting buprenorphine and planning on opioid abstinence

Exclusion Criteria:

1. Pregnant, breast-feeding, or planning on getting pregnant.
2. Alcohol or sedative/hypnotic use disorders (seizure risk).
3. History of/or current psychotic disorder (e.g. schizophrenia).
4. Current or lifetime bipolar disorder.
5. Unstable Axis-I condition requiring starting a new medication.
6. Active suicidal ideation / suicide attempt within 90 days.
7. History of/or current dementia or other cognitive impairment.
8. Contraindications to receiving rTMS or undergoing MRI (implanted ferromagnetic metal, history of or high risk of seizure, implanted device).
9. Unstable general medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Relapse Free survival | Up to 12 weeks
  The number of participants who have not met relapse criteria in the 12-week follow-up phase. Relapse is defined as a) any opioid use in 4 consecutive weeks, or b) any opioid use on 7 consecutive days.

SECONDARY OUTCOMES:
Weeks of opioid abstinance | 12-weeks
  Number of weeks in the 12-week follow-up period that the participant is abstinent from opioids based on self-report and a negative urine drug test

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No